CLINICAL TRIAL: NCT03198585
Title: Empagliflozin in Heart Failure Patients With Reduced Ejection Fraction: A Randomized Clinical Trial (Empire HF)
Brief Title: Empagliflozin in Heart Failure Patients With Reduced Ejection Fraction
Acronym: Empire HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morten Schou (Other)
Responsible Party: Sponsor-Investigator, Morten Schou, MD, PhD, Consultant Cardiologist, Associate Professor, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Empire HF; 2017-001341-27 (EudraCT Number)
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin 10 mg (Active Comparator)
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Capsule, once a day for 90 days
  Arms: Empagliflozin 10 mg
Other: Placebo — Capsule, once a day for 90 days
  Arms: Placebo

SUMMARY:
To assess the effect of Empagliflozin on cardiac biomarkers, cardiac function at rest and during stress, cardiac hemodynamics, renal function, metabolism, daily activity level and health-related quality of life in stable, symptomatic heart failure patients with reduced left ventricular ejection fraction.

The primary hypothesis is that 3 months' treatment with Empagliflozin 10 mg a day will reduce the plasma concentrations of N-terminal pro-brain natriuretic peptide (NT-proBNP).

ELIGIBILITY:
Inclusion Criteria:

* Optimal Heart Failure Therapy in accordance with European and National Guidelines
* LVEF ≤ 0.40
* eGFR > 30 ml/min/1.73 m2
* BMI < 45 kg/m2
* NYHA class I-III
* Age > 18 years
* If T2D - optimal treatment in accordance with European and National Guidelines
* If T2D - stable doses of antiglycemic treatment for 30 days
* If T2D - HbA1C 6.5-10%

Exclusion Criteria:

* CRT-D/-P implanted < 90 days
* Uncorrected severe valvular disease
* Non-compliance
* Use of metalozone
* NYHA IV
* Age > 85 years
* Dementia
* Admission for HF < 30 days
* Admission for hypoglycemia < 12 month
* Known sustained VT
* Symptomatic hypotension and systolic BP < 95 mmHg
* Unable to perform an exercise test
* Immobilization
* Pregnancy
* Participation in other medical trials
* Previous intolerance of Empagliflozin or excipients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Between-group difference in the change of plasma concentrations of NT-proBNP | 90 days

SECONDARY OUTCOMES:
Between-group difference in the change in daily activity level measured by patient-worn accelerometers as change in the amount of daily average accelerometer units | 90 days
Between-group difference in the change in body composition assessed by DXA scan | 90 days
Between-group difference in the change of estimated extracellular volume assessed by Cr-51 EDTA clearance | 90 days
Between-group difference in the change of estimated plasma volume assessed by hematocrit and hemoglobin | 90 days
Between-group difference in the change of glucose metabolism assessed by oral glucose tolerance test | 90 days
Between-group difference in the change of ketone supply to the heart assessed by blood ketones | 90 days
Between-group difference in the change of renal function assessed by Cr-51 EDTA clearance | 90 days
Between-group difference in the change of uric acid | 90 days
Between-group difference in the change of urine albumin/creatinine ratio | 90 days
Between-group difference in the change of cardiac biomarkers assessed by plasma concentrations of MR-proADM and hs-cTnI | 90 days
Between-group difference in the change of cardiac systolic and diastolic function including left ventricular global longitudinal strain and left ventricular ejection fraction assessed by transthoracic echocardiography at rest and during stress | 90 days
Between-group difference in the change of cardiac hemodynamics during rest and sub-maximal exercise assessed by right heart catheterization including pulmonary capillary wedge pressure to cardiac index ratio | 90 days
Between-group difference in the change of cardiac hemodynamics during rest and sub-maximal exercise assessed by right heart catheterization including left ventricular contractile reserve | 90 days
Between-group difference in the change of health-related quality of life assessed by the questionnaire KCCQ | 90 days
Between-group difference in the change of health-related quality of life assessed by the questionnaire EQ-5D-5L | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Morten Schou, MD, Principal Investigator — Herlev and Gentofte University Hospital; Jacob E Moller, MD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Herlev and Gentofte University Hospital, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omar M, Jensen J, Frederiksen PH, Ali M, Kistorp C, Videbaek L, Poulsen MK, Tuxen CD, Borlaug BA, Moller S, Gustafsson F, Kober L, Schou M, Moller JE. Effects of Empagliflozin on Right Ventricular Function in Heart Failure with Reduced Ejection Fraction. medRxiv [Preprint]. 2025 Jun 2:2025.05.30.25328686. doi: 10.1101/2025.05.30.25328686. PMID 40502611
- [Derived] Jensen J, Omar M, Kistorp C, Tuxen C, Poulsen MK, Faber J, Kober L, Gustafsson F, Moller JE, Schou M. Effect of Empagliflozin on Multiple Biomarkers in Heart Failure: Insights From the Empire Heart Failure Trial. Circ Heart Fail. 2022 Aug;15(8):e009333. doi: 10.1161/CIRCHEARTFAILURE.121.009333. Epub 2022 Apr 21. No abstract available. PMID 35973031
- [Derived] Omar M, Jensen J, Kistorp C, Hojlund K, Videbaek L, Tuxen C, Larsen JH, Andersen CF, Gustafsson F, Kober L, Schou M, Moller JE. The effect of empagliflozin on growth differentiation factor 15 in patients with heart failure: a randomized controlled trial (Empire HF Biomarker). Cardiovasc Diabetol. 2022 Feb 27;21(1):34. doi: 10.1186/s12933-022-01463-2. PMID 35219331
- [Derived] Omar M, Jensen J, Burkhoff D, Frederiksen PH, Kistorp C, Videbaek L, Poulsen MK, Gustafsson F, Kober L, Borlaug BA, Schou M, Moller JE. Effect of Empagliflozin on Blood Volume Redistribution in Patients With Chronic Heart Failure and Reduced Ejection Fraction: An Analysis From the Empire HF Randomized Clinical Trial. Circ Heart Fail. 2022 Mar;15(3):e009156. doi: 10.1161/CIRCHEARTFAILURE.121.009156. Epub 2021 Nov 8. PMID 34743533
- [Derived] Omar M, Jensen J, Frederiksen PH, Videbaek L, Poulsen MK, Brond JC, Gustafsson F, Borlaug BA, Schou M, Moller JE. Hemodynamic Determinants of Activity Measured by Accelerometer in Patients With Stable Heart Failure. JACC Heart Fail. 2021 Nov;9(11):824-835. doi: 10.1016/j.jchf.2021.05.013. Epub 2021 Sep 8. PMID 34509409
- [Derived] Jensen J, Omar M, Kistorp C, Tuxen C, Gustafsson I, Kober L, Gustafsson F, Faber J, Forman JL, Moller JE, Schou M. Metabolic Effects of Empagliflozin in Heart Failure: A Randomized, Double-Blind, and Placebo-Controlled Trial (Empire HF Metabolic). Circulation. 2021 Jun;143(22):2208-2210. doi: 10.1161/CIRCULATIONAHA.120.053463. Epub 2021 Jun 1. No abstract available. PMID 34061581
- [Derived] Omar M, Jensen J, Ali M, Frederiksen PH, Kistorp C, Videbaek L, Poulsen MK, Tuxen CD, Moller S, Gustafsson F, Kober L, Schou M, Moller JE. Associations of Empagliflozin With Left Ventricular Volumes, Mass, and Function in Patients With Heart Failure and Reduced Ejection Fraction: A Substudy of the Empire HF Randomized Clinical Trial. JAMA Cardiol. 2021 Jul 1;6(7):836-840. doi: 10.1001/jamacardio.2020.6827. PMID 33404637
- [Derived] Jensen J, Omar M, Kistorp C, Tuxen C, Gustafsson I, Kober L, Gustafsson F, Faber J, Malik ME, Fosbol EL, Bruun NE, Forman JL, Jensen LT, Moller JE, Schou M. Effects of empagliflozin on estimated extracellular volume, estimated plasma volume, and measured glomerular filtration rate in patients with heart failure (Empire HF Renal): a prespecified substudy of a double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2021 Feb;9(2):106-116. doi: 10.1016/S2213-8587(20)30382-X. Epub 2020 Dec 22. PMID 33357505
- [Derived] Jensen J, Omar M, Kistorp C, Poulsen MK, Tuxen C, Gustafsson I, Kober L, Gustafsson F, Fosbol E, Bruun NE, Videbaek L, Frederiksen PH, Moller JE, Schou M. Empagliflozin in heart failure patients with reduced ejection fraction: a randomized clinical trial (Empire HF). Trials. 2019 Jun 21;20(1):374. doi: 10.1186/s13063-019-3474-5. PMID 31227014